CLINICAL TRIAL: NCT01181258
Title: Lymphodepleting Chemotherapy With Rituximab and Allogeneic Natural Killer Cells for Patients With Refractory Lymphoid Malignancies (MT2009-15)
Brief Title: Penostatin, Rituximab and Ontak and Allogeneic Natural Killer (NK) Cells for Refractory Lymphoid Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009LS083; MT2009-15 (Other: Blood and Marrow Transplantation Program); 1002M77545 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2016-01

CONDITIONS: Non-Hodgkin Lymphoma; Chronic Lymphocytic Leukemia
Keywords: related HLA-haploidentical donor
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Interleukin-2; IL32 protein, human; Cyclophosphamide; Methylprednisolone; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients Receiving NK Cell Infusion (Experimental): Non-Myeloablative Conditioning Using Rituximab, Fludarabine, Cyclophosphamide and Methylprednisolone followed by Interleukin 2-activated Allogeneic Natural Killer Cells infusion for Patients with Refractory NHL and CLL
  Interventions: Drug: Rituximab; Biological: Interleukin-2; Biological: Natural killer cells; Drug: Cyclophosphamide; Drug: Methylprednisolone; Drug: Fludarabine

INTERVENTIONS:
Drug: Rituximab — 375 mg/m^2 administered intravenously (IV) weekly * 4, (day -7, -1, +6, +13) pre-infusion with natural killer cells (NK)
  Other Names: Rituxan; MabThera
Biological: Interleukin-2 — subcutaneously administered 9 million international units (IU) every other day * 6 doses over 2 weeks begin 1 to 24 hours after NK cell infusion. If weight < 45 kilograms, give IL-2 at 5 million units/m2 on same schedule.
  Other Names: IL-2
Biological: Natural killer cells — administered intravenously 1.5 to 8 * 10^7 cells/kg on Day 0 (day of NK cell infusion)
  Other Names: NK cells
Drug: Cyclophosphamide — 60 mg/kg administered intravenously (IV) for 2 hours on day -5 after Fludarabine.
  Other Names: Cytoxan
Drug: Methylprednisolone — 1 mg/kg on Days -2 through +9 as an intravenous (IV) infusion.
  Other Names: Medrol
Drug: Fludarabine — 25 mg/m^2/day administered as a 1 hour IV infusion once a day for 5 doses (day -6 through day -2).
  Other Names: Fludara

SUMMARY:
In this study the investigators investigate a cell therapy strategy that could harness allogeneic effectors that can potentially mediate anti-lymphoma effect. The investigators have designed a novel lymphodepleting conditioning regimen followed by infusion of donor-derived natural killer (NK) cells and interleukin-2 (IL-2) for patients with refractory lymphoid malignancies.

DETAILED DESCRIPTION:
This is a single center phase II trial designated to expand donor NK cells and induce remissions in patients with refractory non-Hodgkin lymphoma (NHL) and chronic lymphocytic leukemia (CLL) using chemotherapy followed by haploidentical NK cells and IL2.

Primary Objective is to evaluate the objective response rate (PR+CR) at 2 months post haploidentical NK cell infusion in patients with refractory Non Hodgkin's Lymphoma (NHL) and chronic lymphocytic leukemia (CLL).

Secondary Objective is to 1) evaluate the safety and tolerability of lymphodepleting chemotherapy, rituximab, and methylprednisone as determined by incidence of serious adverse events; 2) evaluate in vivo expansion of allogeneic donor NK cells at day 14; 3) determine time to progression

Exploratory Objective is to 1) correlate clinical response with frequencies of peripheral blood T reg cells after chemotherapy; 2) correlate clinical response with donor KIR-B-content score determined by genotype; 3) monitor phenotypic and functional characteristics of natural killer cells and regulatory T cells in vivo; 4) correlate clinical response with donor FcR polymorphism.

* Pre-NK cell infusion chemotherapeutic regimen consist of 1) Rituximab 375mg/m2 IV weekly x 4, start day -7; 2) Fludarabine 25 mg/m2 IV day -6 through day -2; 3) Cyclophosphamide 60mg/kg IV day -5; 4) Methylprednisolone 1 mg/kg day -2 through day +9.
* NK cell infusion using IL2 activated donor NK cells 1.5 to 8 x 107 cells/kg IV day 0
* IL2 SC 9 million IU every other day x 6 doses over 2 weeks begin 1 to 24 hours after NK cell infusion. If weight < 45 kilograms, give IL-2 at 5 million units/m2 on same schedule

Accrual Goal: Up to 17 patients will be enrolled

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age with diagnosis of:

  * Relapsed/refractory lymphoma (B cell non-Hodgkin) who have lack of objective response to at least two prior chemotherapy regimens
  * Relapsed chronic lymphocytic leukemia with high risk features: lack of objective response or relapse within 6 months following nucleoside-analogue based chemotherapy regimen or patients with 17p deletion CLL who lacked objective response to at least 1 preceding chemotherapy regimen
* Available related HLA haploidentical NK cell donor by at least Class I serologic typing at the A&B locus (age 12-75 years)
* Karnofsky > 70% for patients 16 years and older and Lansky play score > 50 for patients under 16 years of age
* Measurable disease based on modified Response Evaluation Criteria in Solid Tumors (RECIST)
* Have acceptable organ function as defined within 28 days of enrollment:

  * Hematologic: platelets ≥ 80,000 x 10^9/L; hemoglobin ≥ 9 g/dL, unsupported by transfusions within 7 days; absolute neutrophile count (ANC) ≥ 1000 x 10^9/L, unsupported by Granulocyte colony-stimulating factor (G-CSF) or Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) for 10 days or Neulasta for 21 days - the hematologic requirements are waived for patients with inadequate counts due to known bone marrow involvement by disease who are otherwise eligible
  * Renal: calculated glomerular filtration rate (GFR) > 50 ml/min
  * Hepatic: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 5 x upper limit of normal and total bilirubin ≤3 mg/dl - hepatic requirements are waived for patients with known disease involvement in the liver if otherwise eligible
  * Pulmonary function: >40% corrected Carbon Monoxide Diffusing Capacity (DLCO) and Forced expiratory volume in one second (FEV1) (oxygen saturation [>92%] can be used in child where pulmonary function tests (PFT's) cannot be obtained)
  * Cardiac: no symptoms of uncontrolled cardiac disease, left ventricular ejection fraction ≥ 40%
* Able to be off prednisone or other immunosuppressive medications for at least 3 day prior to Day 0 (excluding denileukin diftitox pre-medications)
* Sexually active women of childbearing potential must agree to use adequate contraception (diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.) for the duration of treatment.
* Voluntary written consent

Exclusion Criteria:

* Pregnant or lactating. The agents used in this study may be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. All females of childbearing potential must have a blood test or urine study within 14 days prior to enrollment to rule out pregnancy. Women of childbearing age must use appropriate contraceptive method.
* Active central nervous system (CNS) lymphoma/leukemia - Patients with prior CNS involvement are eligible provided that it has been treated and is in remission.
* Active serious infection (pulmonary infiltrates or lesions are allowed only after the appropriate diagnostic testing is negative for infection or appropriate therapy was initiated for probable infection)
* Pleural effusion large enough to be detectable on chest x-ray (CXR)
* Evidence of human immunodeficiency virus (HIV) infection or known HIV positive serology
* Active concurrent malignancy (except skin cancer)
* Epstein-Barr virus (EBV) post-transplant lymphoproliferative disorder
* Positive HBsAg. If HBcAb is positive, Hepatitis B DNA by PCR will be evaluated. Positive anti HBcAb with an undetectable viral load does not exclude the patient.
* Any investigational therapy in the past 30 days
* Patients following allogeneic stem cell transplantation are eligible in the absence of graft versus host disease and are off immunosuppression for at least 30 days
* Known allergy to any of the study agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-08; Primary Completion 2015-09 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Bachanova, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Bachanova V, Sarhan D, DeFor TE, Cooley S, Panoskaltsis-Mortari A, Blazar BR, Curtsinger JM, Burns L, Weisdorf DJ, Miller JS. Haploidentical natural killer cells induce remissions in non-Hodgkin lymphoma patients with low levels of immune-suppressor cells. Cancer Immunol Immunother. 2018 Mar;67(3):483-494. doi: 10.1007/s00262-017-2100-1. Epub 2017 Dec 7. PMID 29218366

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Receiving NK Cell Infusion: Non-Myeloablative Conditioning Using Rituximab, Fludarabine, Cyclophosphamide and Methylprednisolone followed by Interleukin 2-activated Allogeneic Natural Killer Cells infusion for Patients with Refractory NHL and CLL
  Rituximab: 375 mg/m^2 administered intravenously (IV) weekly * 4, (day -7, -1, +6, +13) pre-infusion with natural killer cells (NK)
  Interleukin-2: subcutaneously administered 9 million international units (IU) every other day * 6 doses over 2 weeks begin 1 to 24 hours after NK cell infusion. If weight < 45 kilograms, give IL-2 at 5 million units/m2 on same schedule.
  Natural killer cells: administered intravenously 1.5 to 8 * 10^7 cells/kg on Day 0 (day of NK cell infusion)
  Cyclophosphamide: 60 mg/kg administered intravenously (IV) for 2 hours on day -5 after Fludarabine
  Methylprednisolone: 1 mg/kg on Days -2 through +9 as an intravenous (IV) infusion
  Fludarabine: 25 mg/m^2/day administered as a 1 hour IV infusion once a day for 5 doses (day -6 through
Period: Overall Study
Arm/Group | Patients Receiving NK Cell Infusion
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Receiving NK Cell Infusion
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With an Objective Response
Description: The number of patients with a partial response (PR) or complete response (CR). For patients with non-hodgkin's lymphoma: CR - complete disappearance of all detectable clinical evidence of disease and disease-related symptoms. PR - at least a 50% decrease in sum of the product of the diameters of up to six of the largest dominant nodes or nodal masses. For patients with chronic lymphocytic leukemia: CR - disappearance of all palpable disease, normalization of the blood counts without transfusions, bone marrow aspirate lymphocyte percentage < 30%, and no evidence of disease on bone marrow biopsy. PR - 50% or more reduction in palpable disease as well as one or more of the remaining features: neutrophils >= 1.5 × 109/L or 50% improvement over baseline, platelets more than 100 × 109/L or 50% improvement over baseline, and hemoglobin more than 11.0 g/dL or 50% improvement over baseline without transfusions.
Time Frame: Month 2 Post Infusion
Population: Two participants were not evaluable. One patient died prior to receiving NK cell infusion and one did not survive by day 14; therefore 14 patients were analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Receiving NK Cell Infusion
Number analyzed (Participants) | 14
Participants | 4

2. Secondary Outcome: Serious Adverse Events
Description: Number of participants experiencing serious adverse events that occur during study. Adverse event collection for the purposes of this study will focus on targeted adverse events and unexpected adverse events at specific time points in relation to the NK cell infusion and post infusion IL2 injections.
Time Frame: Day 1 through Month 12
Population: One participant developed sepsis prior to receiving the NK cell infusion and was withdrawn from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Receiving NK Cell Infusion
Number analyzed (Participants) | 15
Participants | 15

3. Secondary Outcome: Time to Disease Progression
Description: Cumulative incidence will be used to determine time to disease progression.
Time Frame: Day 1 through Month 12
Population: 10 participants had disease progression
Measure: Median (Full Range); unit: days
Arm/Group | Patients Receiving NK Cell Infusion
Number analyzed (Participants) | 10
days | 38 [22 to 43]

4. Secondary Outcome: Patients With Expansion of NK Cells
Description: Number of patients who experience in vivo expansion of allogeneic donor natural killer (NK) cells.
Time Frame: Day 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Receiving NK Cell Infusion
Number analyzed (Participants) | 14
Participants | 0

ADVERSE EVENTS:
Description: Fifteen patients were dosed with the NK cell infusion and therefore were assessed for adverse events. One patient died prior to the NK cell infusion.
Arm/Group | Patients Receiving NK Cell Infusion
Serious Adverse Events (participants affected / at risk) | 6/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Receiving NK Cell Infusion (N=15)
Sepsis (Infections and infestations) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Cardiac disorders) | 1
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Receiving NK Cell Infusion (N=15)
Acute Kidney Injury (Renal and urinary disorders) | 2
Back/Chest Spasms (Musculoskeletal and connective tissue disorders) | 1
Capillary Leak Syndrome (Vascular disorders) | 1
Chemosis, Eye (Eye disorders) | 1
Chest Pain (General disorders) | 1
Chills (General disorders) | 14
Confusion (Psychiatric disorders) | 1
Creatinine Increased (Investigations) | 3
Dry Eyes (Eye disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Edema (General disorders) | 8
Fever (General disorders) | 9
Flu-like Symptoms (General disorders) | 1
Headache (Nervous system disorders) | 6
Hypertension (Vascular disorders) | 14
Hypotension (Vascular disorders) | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Infusion Related Reaction (General disorders) | 6
Injection Site Reaction (General disorders) | 8
Left Jaw Pain (Musculoskeletal and connective tissue disorders) | 1
Leg Pain (Musculoskeletal and connective tissue disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Neutropenic Fever (Blood and lymphatic system disorders) | 8
Peripheral Neuropathy (Nervous system disorders) | 1
Pneumonitis/Pulmonary Infiltrates (Respiratory, thoracic and mediastinal disorders) | 3
Prolonged QTC Interval (Cardiac disorders) | 1
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 7
Tachycardia (Cardiac disorders) | 2
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1
Tumor Pain (General disorders) | 1
Upper Extremity Swelling/Edema (General disorders) | 2
Weight Gain (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No